CLINICAL TRIAL: NCT04844099
Title: Dihydroartemisinin-Piperaquine or Sulphadoxine-Pyrimethamine for the Chemoprevention of Malaria in Children With Sickle Cell Anaemia in Eastern and Southern Africa: a Double Blind Randomised Trial (CHEMCHA)
Brief Title: Dihydroartemisinin-Piperaquine or Sulphadoxine-Pyrimethamine for the Chemoprevention of Malaria in Sickle Cell Anaemia
Acronym: CHEMCHA
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: University of Bergen (Other); University of Malawi (Other); Makerere University (Other); Indiana University (Other); Global Health Uganda LTD (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 19-105
Record Dates: First submitted 2021-03-26; First posted 2021-04-14 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2022-09

CONDITIONS: Sickle Cell Anemia in Children; Malaria
Keywords: dihydroartemisinin-piperaquine; sulphadoxine pyrimethamine; sickle cell; malaria; chemoprevention; prophylaxis
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Intervention Model Description: This will be a randomized, double-blind, parallel-group superiority trial of weekly single-day courses of DP for an average of 18 months compared to monthly single-day courses of SP in SCA patients. The study will be conducted in Uganda and Malawi, using randomisation stratified by bodyweight and study centre. Participants will be randomized using an allocation of 1:1 to DP or SP. Patients on DP will also receive an SP placebo, and those on SP will in addition, receive a DP placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This will be a double-blinded study. Patients on DP will also receive SP placebo, and those on SP will in addition, receive DP placebo. All laboratory staff will be masked to the treatment assignment of individual participants. The trial statistician will also be blinded regarding the treatment code when he/she develops the statistical analysis plan and writes the statistical programmes, which will be validated and completed using dummy randomisation codes.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): The intervention will be oral dihydroartemisinin (20mg) and piperaquine (160 mg) and administered once weekly at approximate doses of dihydroartemisinin 2.5mg/kg/day and piperaquine 20mg/kg/day based on participants' weight categories
  Interventions: Drug: Dihydroartemisinin Piperaquine
- Comparator (Active Comparator): The active control will be Sulphadoxine-Pyrimethamine (SP), the current standard of care for malaria chemoprevention for SCA in Uganda and Malawi. This will also be provided by Guilin Pharmaceutical Co. Ltd as their generic World Health Organization-approved sulphadoxine-pyrimethamine 500/25mg tablets. It will be administered as monthly single-day courses of SP at approximate doses of S=25mg/kg and P=1.25mg/kg.
  Interventions: Drug: Dihydroartemisinin Piperaquine

INTERVENTIONS:
Drug: Dihydroartemisinin Piperaquine — Administered as dihydroartemisinin (20mg) and piperaquine (160 mg)
  Other Names: D-ARTEPP® (Guilin Pharmaceutical Co. Ltd)

SUMMARY:
Sickle Cell Anaemia (SCA) is an inherited disease that makes the body produce red blood cells with abnormal sickle-shaped cells. The sickle-shaped cells are rigid, not flexible and break up easily resulting in anaemia. The abnormal cells also stick to the vessel walls, causing a blockage that slows or stops the flow of blood. When this happens, oxygen cannot reach nearby tissues. The lack of oxygen can cause attacks of sudden, severe pain, called pain crises, stroke or damage to important organs such as the spleen. All of these can lead to death. These attacks can occur without warning and are often started and made worse by infections such as malaria. Therefore, in many countries in Africa where malaria is common, children with SCA are given malaria medicines to prevent the infection. However, many of the medicines do not work effectively, are too difficult to take or they have side effects, resulting in poor adherence.

The aim of this study is to find safe, acceptable and effective medicines for malaria prevention in children with SCA in eastern and southern Africa. The investigators propose to conduct a study to find out whether giving weekly doses of dihydroartemisinin-piperaquine, also called DP, is safe, more effective, acceptable and cost-effective than the current strategy of monthly sulphadoxine-pyrimethamine (SP) to prevent malaria in children with sickle cell anaemia. Overall, 548 children aged 6 months to 15 years will be chosen randomly to receive either weekly DP or monthly SP for about 18 months. To test if the study medicine is effective, the study will compare the case burden of malaria. The investigators will also monitor every child for any type of illness, blood transfusions and other complications of sickle cell anaemia and admissions to the hospital. In addition, the study will evaluate the impact of DP on the development of resistance by malaria parasites. The study will also include nested safety studies on the effect of DP on the heart. All study participants will receive all the other usual care and treatments, including patient education on home care, and daily penicillin if younger than 5 years. If proven safe and efficacious, chemoprophylaxis with DP may decrease the incidence of malaria in children with SCA, prevent ill-health and deaths, and improve wellbeing.

DETAILED DESCRIPTION:
Background and rationale:

An estimated 300,000 babies are born with Sickle Cell Anaemia (SCA) annually. Affected children have chronic ill health and many suffer a premature death. Ill health is commonly precipitated by febrile illnesses including malaria. Antimalarial chemoprophylaxis is an important strategy, but current regimes are either sub-optimally effective (e.g., monthly sulphadoxine-pyrimethamine, SP) or difficult to adhere to (e.g., daily proguanil). The investigators propose dihydroartemisinin-piperaquine (DP) as the agent with the most potential to be used across Africa.

Objectives:

Our objective is to determine the efficacy, safety, uptake, and cost-effectiveness of malaria chemoprevention with weekly single day courses of DP vs monthly single day courses of SP in children with SCA in eastern and southern Africa.

Hypothesis:

The hypothesis is that weekly single day courses of DP, is safe and more efficacious, compared to monthly single day courses of SP, for the malaria chemoprevention in children with SCA in eastern and southern Africa.

Design:

This will a randomised, double-blind controlled parallel-group superiority trial of weekly single day courses of DP for an average of 18 months compared to monthly single-day courses of SP in SCA patients. The study will be conducted in Uganda and Malawi. Participants will be randomised to DP or SP (1:1), stratified by bodyweight and study centre. The study will also assess the acceptability and uptake of the two interventions, the safety and pharmacokinetics of weekly DP, the development of resistance to DP and cost-effectiveness. At the end of the study, this information will be used to inform regional health policy.

Sites:

Participants will be recruited from Jinja Regional Referral hospital and Kitgum General hospital in Uganda and Queen Elizabeth (Blantyre) hospital in Malawi.

Interventions:

The intervention will be oral DP administered weekly for an average of 18 months based on weight categories. DP will be provided as tablets of D-ARTEPP® (Guilin Pharmaceutical Co. Ltd) and administered as dihydroartemisinin (20mg) and piperaquine (160 mg) at approximate doses of dihydroartemisinin 2.5mg/kg/day and piperaquine 20mg/kg/day. The active control will be the current standard of care for chemoprevention in Uganda and Malawi - monthly single-dose SP (S=25mg/kg). The same manufacturer will provide SP as the generic SP (in 500/25mg scored tablets).

Other care:

In addition to the above-mentioned malaria regimens, the participants will receive the standard of care for Sickle Cell Anaemia (including parental education on care, treatment for both the acute and chronic complications of Sickle Cell Anaemia, and daily penicillin prophylaxis if <5 years).

Sample size:

With the minimum incidence rate of clinical malaria in SCA patients receiving monthly SP estimated at 0.2 events per year, and an effect size of 50% if DP is used, at a power of 0.9 and 0.05 level of significance, followed up for 18 months and allowing for 20% losses to follow up, and one interim analysis, the investigators will need 548 participants (274 in either arm) followed up for an average 18 months or until 824 person-years.

Follow up:

Participants will be followed for up for an average of 18 months or until 412 person-years of observation is achieved in each group (a combined total of 824 person-years of observation). This will be achieved by following between 548 and 824 participants for an average of 12 to 18 months each.

Outcome measures:

The primary efficacy outcome measures will be the incidence of clinical malaria. Secondary efficacy outcomes will include the incidence of malaria parasitaemia, all-cause sick-child clinic visits, SCA-related vaso-occlusive events (including severe pain events and dactylitis), acute chest syndrome, stroke, hospitalisations, blood-transfusions, and death.

Secondary safety outcome measures: QTc-prolongation on ECG recordings and incidence of serious cardiac adverse events (e.g., convulsions or syncope within 48 hours after drug intake). Tolerance: % vomiting drug within 30 minutes of administration. Others are cost-effectiveness, development of resistance to piperaquine, feasibility, acceptability, and uptake.

Data Analysis: Primary analysis will be by intention to treat. Incidence rates will be calculated, and rate ratios estimated using Poisson regression, with treatment (as randomised) as the predictor variable and the stratification factors site and weight-band as covariates.

ELIGIBILITY:
Inclusion criteria

1. Children ages 6 months - 15 years
2. Has a laboratory diagnosis of Sickle Cell Anaemia (HbSS) on haemoglobin electrophoresis, High-Performance Liquid Chromatography or Iso-electric focusing;
3. Weighs ≥5kg;
4. The parent has provided written consent.

Exclusion Criteria:

1. Known chronic disease e.g. congenital heart disease;
2. Known red cell disorder e.g. thalassaemia, glucose-6-phosphate dehydrogenase deficiency;
3. Known allergy to DP or SP;
4. Receiving daily cotrimoxazole prophylaxis;
5. Unlikely to comply with the follow-up schedule;
6. Participating in another trial

Ages: 6 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 723 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
Incidence of clinical malaria | 18 months
  An episode of malaria will be defined as a history of fever in the preceding 48hrs or documented axillary temperature ≥37.5 degrees centigrade plus microscopy confirmed Plasmodium falciparum malaria

SECONDARY OUTCOMES:
All cause sick visits | 18 months
  The incidence of all cause sick visits
Incidence of malaria parasitaemia | 18 months
  The incidence of malaria parasitaemia
Malaria specific sick visits | 18 months
  The incidence of malaria-specific sick visits
All-cause and malaria-specific hospitalisation | 18 months
  The incidence of all-cause and malaria-specific hospitalisation
Sickle Cell Anaemia-related vaso-occlusive events | 18 months
  The incidence of SCA-related vaso-occlusive events (including severe pain events and dactylitis); acute chest syndrome, stroke and need for blood transfusion
Death | 18 months
  The incidence of death.
QTc prolongation | 18 months
  Change in Corrected QT interval (QTc) length and QTc-prolongation on four-monthly ECG recordings.
Serious cardiac adverse events | 18 months
  Incidence of serious cardiac adverse events (e.g., convulsions or syncope within 48 hours after drug intake)
Serious adverse events | 18 months
  Incidence of serious adverse events
Tolerance - vomiting | 18 months
  1. Vomiting the study drug within 30 min of administration;
  2. Incidence of gastrointestinal complaints.
Other gastro-intestinal complaints | 18 months
  Incidence of gastrointestinal complaints.
Level of adherence | 18 months
  Level of adherence to study drugs
Provider costs | 18 months
  Provider costs of delivering the interventions and provider costs of managing malaria in SCA children.
Direct and indirect costs | 18 months
  Direct and indirect costs of patients receiving the interventions and managing cases of malaria.
Incremental cost-effectiveness | 18 months
  Incremental cost-effectiveness of replacing current standards of care (SP) with DP or DP+SP from the perspectives of the health care provider and the society.

CONTACTS AND LOCATIONS:
Overall Officials: Robberstad Bjarne, PhD, Study Director — University of Bergen, Norway
Locations (3):
- Queen Elizabeth Hospital, Blantyre, Malawi
- Uganda (2):
  - Jinja Regional Referral hospital, Jinja
  - Kitgum General Hospital, Kitgum

IPD SHARING:
Plan to Share IPD: Yes
At the end of the study, anonymised data will be available to other researchers for further analysis,
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Beginning of 2025
Access Criteria: 1. Ethical approval has been obtained.
  2. The terms of the original patient consent are not violated.
  3. The agreement on its use is according to prevailing laws on intellectual property rights.

REFERENCES:
- [Background] Weatherall D, Hofman K, Rodgers G, Ruffin J, Hrynkow S. A case for developing North-South partnerships for research in sickle cell disease. Blood. 2005 Feb 1;105(3):921-3. doi: 10.1182/blood-2004-06-2404. Epub 2004 Oct 5. PMID 15466925
- [Background] Eridani S. Sickle cell protection from malaria. Hematol Rep. 2011 Oct 19;3(3):e24. doi: 10.4081/hr.2011.e24. Epub 2011 Nov 4. PMID 23285410
- [Background] McAuley CF, Webb C, Makani J, Macharia A, Uyoga S, Opi DH, Ndila C, Ngatia A, Scott JA, Marsh K, Williams TN. High mortality from Plasmodium falciparum malaria in children living with sickle cell anemia on the coast of Kenya. Blood. 2010 Sep 9;116(10):1663-8. doi: 10.1182/blood-2010-01-265249. Epub 2010 Jun 8. PMID 20530796
- [Background] Sinclair D, Zani B, Donegan S, Olliaro P, Garner P. Artemisinin-based combination therapy for treating uncomplicated malaria. Cochrane Database Syst Rev. 2009 Jul 8;2009(3):CD007483. doi: 10.1002/14651858.CD007483.pub2. PMID 19588433
- [Background] Cisse B, Cairns M, Faye E, NDiaye O, Faye B, Cames C, Cheng Y, NDiaye M, Lo AC, Simondon K, Trape JF, Faye O, NDiaye JL, Gaye O, Greenwood B, Milligan P. Randomized trial of piperaquine with sulfadoxine-pyrimethamine or dihydroartemisinin for malaria intermittent preventive treatment in children. PLoS One. 2009 Sep 28;4(9):e7164. doi: 10.1371/journal.pone.0007164. PMID 19784374
- [Background] Lwin KM, Phyo AP, Tarning J, Hanpithakpong W, Ashley EA, Lee SJ, Cheah P, Singhasivanon P, White NJ, Lindegardh N, Nosten F. Randomized, double-blind, placebo-controlled trial of monthly versus bimonthly dihydroartemisinin-piperaquine chemoprevention in adults at high risk of malaria. Antimicrob Agents Chemother. 2012 Mar;56(3):1571-7. doi: 10.1128/AAC.05877-11. Epub 2012 Jan 17. PMID 22252804
- [Background] Kwambai TK, Dhabangi A, Idro R, Opoka R, Kariuki S, Samuels AM, Desai M, van Hensbroek MB, John CC, Robberstad B, Wang D, Phiri K, Ter Kuile FO. Malaria chemoprevention with monthly dihydroartemisinin-piperaquine for the post-discharge management of severe anaemia in children aged less than 5 years in Uganda and Kenya: study protocol for a multi-centre, two-arm, randomised, placebo-controlled, superiority trial. Trials. 2018 Nov 6;19(1):610. doi: 10.1186/s13063-018-2972-1. PMID 30400934
- [Background] Mytton OT, Ashley EA, Peto L, Price RN, La Y, Hae R, Singhasivanon P, White NJ, Nosten F. Electrocardiographic safety evaluation of dihydroartemisinin piperaquine in the treatment of uncomplicated falciparum malaria. Am J Trop Med Hyg. 2007 Sep;77(3):447-50. PMID 17827358
- [Background] Keating GM. Dihydroartemisinin/Piperaquine: a review of its use in the treatment of uncomplicated Plasmodium falciparum malaria. Drugs. 2012 May 7;72(7):937-61. doi: 10.2165/11203910-000000000-00000. PMID 22515619
- [Background] Gutman J, Kovacs S, Dorsey G, Stergachis A, Ter Kuile FO. Safety, tolerability, and efficacy of repeated doses of dihydroartemisinin-piperaquine for prevention and treatment of malaria: a systematic review and meta-analysis. Lancet Infect Dis. 2017 Feb;17(2):184-193. doi: 10.1016/S1473-3099(16)30378-4. Epub 2016 Nov 17. PMID 27865890
- [Background] O'Meara WP, Breman JG, McKenzie FE. The promise and potential challenges of intermittent preventive treatment for malaria in infants (IPTi). Malar J. 2005 Jul 20;4:33. doi: 10.1186/1475-2875-4-33. PMID 16033653
- [Background] Nakibuuka V, Ndeezi G, Nakiboneka D, Ndugwa CM, Tumwine JK. Presumptive treatment with sulphadoxine-pyrimethamine versus weekly chloroquine for malaria prophylaxis in children with sickle cell anaemia in Uganda: a randomized controlled trial. Malar J. 2009 Oct 24;8:237. doi: 10.1186/1475-2875-8-237. PMID 19852829
- [Background] Jiang T, Chen J, Fu H, Wu K, Yao Y, Eyi JUM, Matesa RA, Obono MMO, Du W, Tan H, Lin M, Li J. High prevalence of Pfdhfr-Pfdhps quadruple mutations associated with sulfadoxine-pyrimethamine resistance in Plasmodium falciparum isolates from Bioko Island, Equatorial Guinea. Malar J. 2019 Mar 26;18(1):101. doi: 10.1186/s12936-019-2734-x. PMID 30914041
- [Background] Staedke SG, Sendagire H, Lamola S, Kamya MR, Dorsey G, Rosenthal PJ. Relationship between age, molecular markers, and response to sulphadoxine-pyrimethamine treatment in Kampala, Uganda. Trop Med Int Health. 2004 May;9(5):624-9. doi: 10.1111/j.1365-3156.2004.01239.x. PMID 15117308
- [Background] McCollum AM, Mueller K, Villegas L, Udhayakumar V, Escalante AA. Common origin and fixation of Plasmodium falciparum dhfr and dhps mutations associated with sulfadoxine-pyrimethamine resistance in a low-transmission area in South America. Antimicrob Agents Chemother. 2007 Jun;51(6):2085-91. doi: 10.1128/AAC.01228-06. Epub 2007 Feb 5. PMID 17283199
- [Background] Lynch C, Pearce R, Pota H, Cox J, Abeku TA, Rwakimari J, Naidoo I, Tibenderana J, Roper C. Emergence of a dhfr mutation conferring high-level drug resistance in Plasmodium falciparum populations from southwest Uganda. J Infect Dis. 2008 Jun 1;197(11):1598-604. doi: 10.1086/587845. PMID 18471065
- [Background] Chandramohan D, Owusu-Agyei S, Carneiro I, Awine T, Amponsa-Achiano K, Mensah N, Jaffar S, Baiden R, Hodgson A, Binka F, Greenwood B. Cluster randomised trial of intermittent preventive treatment for malaria in infants in area of high, seasonal transmission in Ghana. BMJ. 2005 Oct 1;331(7519):727-33. doi: 10.1136/bmj.331.7519.727. PMID 16195288
- [Background] Pearson RD, Hewlett EL. Use of pyrimethamine-sulfadoxine (Fansidar) in prophylaxis against chloroquine-resistant Plasmodium falciparum and Pneumocystis carinii. Ann Intern Med. 1987 May;106(5):714-8. doi: 10.7326/0003-4819-106-5-714. PMID 3551713
- [Background] Matthews JI, Molitor JT, Hunt KK Jr. Pyrimethamine-induced leukopenia and thrombocytopenia in a patient with malaria and tropical sprue: case report. Mil Med. 1973 May;138(5):280-3. No abstract available. PMID 4196454
- [Background] Oniyangi O, Omari AA. Malaria chemoprophylaxis in sickle cell disease. Cochrane Database Syst Rev. 2006 Oct 18;2006(4):CD003489. doi: 10.1002/14651858.CD003489.pub2. PMID 17054173
- [Background] Kamya MR, Kapisi J, Bigira V, Clark TD, Kinara S, Mwangwa F, Muhindo MK, Kakuru A, Aweeka FT, Huang L, Jagannathan P, Achan J, Havlir DV, Rosenthal PJ, Dorsey G. Efficacy and safety of three regimens for the prevention of malaria in young HIV-exposed Ugandan children: a randomized controlled trial. AIDS. 2014 Nov 28;28(18):2701-9. doi: 10.1097/QAD.0000000000000497. PMID 25493596
- [Background] Bigira V, Kapisi J, Clark TD, Kinara S, Mwangwa F, Muhindo MK, Osterbauer B, Aweeka FT, Huang L, Achan J, Havlir DV, Rosenthal PJ, Kamya MR, Dorsey G. Protective efficacy and safety of three antimalarial regimens for the prevention of malaria in young Ugandan children: a randomized controlled trial. PLoS Med. 2014 Aug 5;11(8):e1001689. doi: 10.1371/journal.pmed.1001689. eCollection 2014 Aug. PMID 25093754
- [Background] Eke FU, Anochie I. Effects of pyrimethamine versus proguanil in malarial chemoprophylaxis in children with sickle cell disease: a randomized, placebo-controlled, open-label study. Curr Ther Res Clin Exp. 2003 Sep;64(8):616-25. doi: 10.1016/j.curtheres.2003.09.003. PMID 24944408
- [Derived] Idro R, Nkosi-Gondwe T, Opoka R, Ssenkusu JM, Dennis K, Tsirizani L, Akun P, Rujumba J, Nambatya W, Kamya C, Phiri N, Joanita K, Komata R, Innussa M, Tenywa E, John CC, Tarning J, Denti P, Wasmann RE, Ter Kuile FO, Robberstad B, Phiri KS. Weekly dihydroartemisinin-piperaquine versus monthly sulfadoxine-pyrimethamine for malaria chemoprevention in children with sickle cell anaemia in Uganda and Malawi (CHEMCHA): a randomised, double-blind, placebo-controlled trial. Lancet Infect Dis. 2025 Jun;25(6):643-655. doi: 10.1016/S1473-3099(24)00737-0. Epub 2024 Dec 20. PMID 39718172
- [Derived] Nkosi-Gondwe T, Robberstad B, Opoka R, Kalibbala D, Rujumba J, Galileya LT, Akun P, Nambatya W, Ssenkusu J, TerKuile F, Phiri K, Idro R. Dihydroartemisinin-piperaquine or sulphadoxine-pyrimethamine for the chemoprevention of malaria in children with sickle cell anaemia in eastern and southern Africa (CHEMCHA): a protocol for a multi-centre, two-arm, double-blind, randomised, placebo-controlled superiority trial. Trials. 2023 Apr 5;24(1):257. doi: 10.1186/s13063-023-07274-4. PMID 37016392